CLINICAL TRIAL: NCT06711367
Title: Comparative Evaluation of the Effectiveness of Custom-designed Dental Storybook Vs Tell Show Do on the Dental Anxiety and Behavior of Children: a Randomized Controlled Trial
Brief Title: Evaluation of Custom-designed Dental Storybook on the Dental Anxiety and Behavior of Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Ibrahim Ezz, Associate professor, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC-D
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Child Behavior; Dental Anxiety
Keywords: dental storybook; tell show do; dental anxiety
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tell show do behavior management technique (Active Comparator)
  Interventions: Behavioral: tell show do behavior management technique
- a costume-designed dental storybook (Experimental)
  Interventions: Behavioral: a costume-designed storybook

INTERVENTIONS:
Behavioral: tell show do behavior management technique — tell show do behavior management technique about the the diagnosis and procedures of dental restoration
  Arms: tell show do behavior management technique
Behavioral: a costume-designed storybook — a costume-designed storybook explaining the diagnosis and procedures of dental restoration
  Arms: a costume-designed dental storybook

SUMMARY:
Conventional behavior management techniques, namely: verbal communication and tell-show-do were used in the operatory for the participating children (Group A). The children allocated in intervention group (Group B) received a costume-designed storybook explaining the diagnosis and procedures of occlusal composite restoration

ELIGIBILITY:
Inclusion Criteria:

* • Healthy children and children/parents can read and understand Arabic.

  * The child needs an occlusal composite restoration.

Exclusion Criteria:

* Children with special needs; children with a complete audiovisual impairment; children with
* Learning difficulties or mental retardation.
* Children who are not Arabic speakers.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Child anxiety | through study completion, an average of four months
  Venham anxiety scale (score from 1-8)

SECONDARY OUTCOMES:
Pulse rate | through study completion, an average of four months
  Pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- October University of Modern Sciences and Arts, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided